CLINICAL TRIAL: NCT03502538
Title: A Comparative Study of the Efficacy in Plaque Removal of Two Manual Toothbrushes Models: Curaprox® CS 5460 Ultra Soft and Oral-B® Indicator Plus
Brief Title: A Comparative Study of the Efficacy in Plaque Removal of Two Manual Toothbrushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Thais Cristina de Souza Alves, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CURAPROX5460-INDICATORPLUS
Record Dates: First submitted 2017-01-29; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Tooth Caries; Dental Plaque
MeSH Terms: conditions — Dental Caries; Dental Plaque

STUDY DESIGN:
Intervention Model Description: This is a study designed where all the participants will have to try the two devices that were being tested.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curaprox 5460 Ultra Soft (Experimental): Brushing with a Curaprox Ultra Soft 5460 toothbrush for one minute timed without orientations about brushing techniques and without supervision
  Interventions: Device: Curaprox 5460 Ultra Soft; Device: Oral-B Indicator Plus
- Oral-B Indicator Plus (Active Comparator): Brushing with a Oral-B Indicator Plus toothbrush for one minute timed without orientations about brushing techniques and without supervision
  Interventions: Device: Curaprox 5460 Ultra Soft; Device: Oral-B Indicator Plus

INTERVENTIONS:
Device: Curaprox 5460 Ultra Soft — The toothbrush Curaprox 5460 Ultra Soft will be the tested toothbrush model, in order to asses its efficacy in plaque removal. Therefore, the study participants should brush their teeth using this toothbrush model, following the instructions of the investigator. From the data collect related in plaque removal the results will be arrived at.
Device: Oral-B Indicator Plus — Following the same method of the Curaprox group intervention, the participants should brush their teeth using the Oral-B Indicator Plus toothbrush and based on the data collect, the results will be compared with the first group of intervention.

SUMMARY:
Objective: To compare the efficacy of Curaprox® CS 5460 Ultra Soft and Oral-B® Indicator Plus toothbrushes in dental plaque removal. Methods: 50 adult participants will be included in the sample. For a period of 24 hours (at two different times), they will be instructed to stop oral hygiene. During the final 4 hours, the interruption of consumption of foods and liquids will be recommended, and in smokers' case, the use of cigarettes. In two clinical visits (T0 and T1), volunteers will be asked to brush their teeth for 1 minute with Curaprox® (CS 5460 Ultra Soft) e Oral-B® (Indicator Plus) toothbrushes. Disclosure will be performed prior to and after brushing and the presence of plaque on the tooth surfaces will be evaluated. Turesky Modified Quigley Hein Plaque Index will be used for the plaque record. For statistical analysis, paired t tests will be performed to compare the effectiveness of toothbrushes and correlation test to assess whether the fact that the patient was aware of the toothbrush that will be used influenced in their performance.

DETAILED DESCRIPTION:
For the study, 50 patients, between 18 and 55 years of age, of both sexes and healthy will be selected. For the study performance, volunteers will be instructed to stop their brushing for 23 to 25 hours before the first clinical visit. In addition, they will be also instructed to stop eating (solid foods and liquids) and to stop the use of cigarettes, if smoker, for 4 hours before evaluation. Prior to the study, a pilot study will be conducted at the University Hospital of Brasília for the researcher calibration using the Turesky Modified Quigley Hein Plaque Index, following the predetermined protocol.

A double-blind crossover study will be designed in which each volunteer will test two different models of toothbrushes. Prior to the beginning of the study, the brushes handle will be hidden with tape in a way that it will be not possible to see the toothbrush trademark. During the two visits, both brushes will be placed on the workbench and in the absence of the researcher, the participant will select one of the brushes. In the following visit, the same procedure will be performed and the participant will use the second brush. A period of washout of at least one week between the the first visit and the second visit will be done to obtain non-interference between results. No brush restriction will be imposed for the participant during this period.

ELIGIBILITY:
Inclusion Criteria:

* Good oral health
* At least, 24 health teeth

Exclusion Criteria:

* Those with any limitations that make it difficult for the dental examination or the performance of brushing, which use removable prostheses, orthodontic appliances, and/or that have malocclusions, and the presence of a gingival recess equal to or greater than 2mm

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Comparison of dental plaque removal between the toothbrushes Curaprox and Oral-B | Five months
  The participants should stay for 24 hours without toothbrushing. After that, their dental surfaces will be stained, evaluated and the amount of dental plaque will be recorded. The first recording of the dental plaque will be registered and the brushing with each toothbrush model (at two different times, being these at least one week apart) was performed. Then, a second registration will be recorded. The measurement will be perfomed by visual assessment, according to the Plaque Index mentioned before. The index is based on the assessment of six areas of the dental surface; three in the buccal surface (mesio, middle and distobuccal) and three on the palatine / lingual surface following the same order (mesio, medium and disto). For each area a value according to the presence of plaque will be recorded. These values can be from 0 to 5. A statistical analysis will be performed to compare the amount of plaque removing after brushing with each toothbrush model.

IPD SHARING:
Plan to Share IPD: Yes
The results will be published. Consent forms and participant information sheets will explain how data will be shared after the study.
Supporting Information: CSR
Time Frame: Data will be available when the journal accept the paper for publication.
Access Criteria: The results will be provided by statistical analysis.